CLINICAL TRIAL: NCT00915148
Title: First Stage 3D-ultrasound During Prolonged Labour.
Brief Title: Ultrasound Prediction of Prolonged Labour
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: StaHF500804
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Prolonged Labor
Keywords: Prolonged labor; Ultrasound; Caeserian section

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound examination: Women with prolonged Labour; Primi gravidae, single pregnancy, >37 weeks, fetus alive, cephalic presentation.
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — Trans-abdominal and trans-perineal 3D ultrasound examination

SUMMARY:
This observational study is designed to correlate findings on ultrasound with manual palpation, and to consider if delivery outcome can be predicted with help of ultrasound. Specifically, the study will evaluate the significance of fetal head level (descent) in the pelvis, measured with ultrasound.

DETAILED DESCRIPTION:
AIM:

To correlate findings on ultrasound with manual palpation, and to consider if delivery outcome can be predicted with help of ultrasound. Specifically evaluate the significance of fetal head level (descent) in the pelvis, measured with ultrasound.

Objective:

Labours have traditionally been evaluated by manuals methods of the "delivery helper" - midwives or doctor. There are many factors that will prolong labour such as malcontractions, disproportion of the birth canal and malpresentation/position. In about 20% of primigravidae, the first stage will last longer than 10 hours.

In this study we want to evaluate different ultrasounds measurements to see if ultrasound can be used to predict the outcome of labour.

Methods:

A descriptive observational study, with one ultrasound examination. The labour will be handled according to definitions by Woman's department, Stavanger University Hospital, and WHO.

The use of stimulating agents, as Oxytocin, will be evaluated after manual examinations, specific definitions and criteria.

The results of the ultrasound examinations will be evaluated after the delivery, since the results are not to be used clinically during the delivery.

Inclusion criteria will be primigravidae, with one fetus, after the 37th week. Feta head presentation. Ruptured membranes, at least one hour before inclusion. Prolonged first stage according to WHO definitions. The target is to include 100 subjects.

Inter- and intraobserver variation will be evaluated with intraclass coefficients. We will analyze operative delivery with normal vaginal delivery. Also, two groups divided by the stage 0 will be evaluated with statistics analyzes.

Time to delivery will be evaluated with Kaplan Meier and Cox regression analyzes.

ELIGIBILITY:
Inclusion Criteria:

* Primi gravidae
* >37th week
* Cephalic presentation
* Prolonged first stage according to WHO definitions.

Exclusion Criteria:

* Multiple pregnancies
* Intrauterine fetal death

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primi gravidae, with one fetus, after the 37th week. Cephalic presentation. Prolonged first stage according to WHO definitions.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Andreas Torkildsen, MD, Principal Investigator — Helse Stavanger HF; Torbjørn Moe Eggebø, MD, PhD, Study Director — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Background] Eggebo TM, Heien C, Okland I, Gjessing LK, Romundstad P, Salvesen KA. Ultrasound assessment of fetal head-perineum distance before induction of labor. Ultrasound Obstet Gynecol. 2008 Aug;32(2):199-204. doi: 10.1002/uog.5360. PMID 18528923
- [Background] Eggebo TM, Heien C, Okland I, Gjessing LK, Smedvig E, Romundstad P, Salvesen KA. Prediction of labour and delivery by ascertaining the fetal head position with transabdominal ultrasound in pregnancies with prelabour rupture of membranes after 37 weeks. Ultraschall Med. 2008 Apr;29(2):179-83. doi: 10.1055/s-2007-963017. Epub 2007 Jun 28. PMID 17599279
- [Background] Eggebo TM, Gjessing LK, Heien C, Smedvig E, Okland I, Romundstad P, Salvesen KA. Prediction of labor and delivery by transperineal ultrasound in pregnancies with prelabor rupture of membranes at term. Ultrasound Obstet Gynecol. 2006 Apr;27(4):387-91. doi: 10.1002/uog.2744. PMID 16565994
- [Background] Barbera AF, Pombar X, Perugino G, Lezotte DC, Hobbins JC. A new method to assess fetal head descent in labor with transperineal ultrasound. Ultrasound Obstet Gynecol. 2009 Mar;33(3):313-9. doi: 10.1002/uog.6329. PMID 19248000
- [Background] Henrich W, Dudenhausen J, Fuchs I, Kamena A, Tutschek B. Intrapartum translabial ultrasound (ITU): sonographic landmarks and correlation with successful vacuum extraction. Ultrasound Obstet Gynecol. 2006 Nov;28(6):753-60. doi: 10.1002/uog.3848. PMID 17063455
- [Result] Torkildsen EA, Salvesen KA, Eggebo TM. Prediction of delivery mode with transperineal ultrasound in women with prolonged first stage of labor. Ultrasound Obstet Gynecol. 2011 Jun;37(6):702-8. doi: 10.1002/uog.8951. Epub 2011 May 3. PMID 21308837
- [Result] Tutschek B, Torkildsen EA, Eggebo TM. Comparison between ultrasound parameters and clinical examination to assess fetal head station in labor. Ultrasound Obstet Gynecol. 2013 Apr;41(4):425-9. doi: 10.1002/uog.12422. Epub 2013 Mar 14. PMID 23371409
- [Result] Torkildsen EA, Salvesen KA, Eggebo TM. Agreement between two- and three-dimensional transperineal ultrasound methods in assessing fetal head descent in the first stage of labor. Ultrasound Obstet Gynecol. 2012 Mar;39(3):310-5. doi: 10.1002/uog.9065. PMID 21630362

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical contact during10 months
Pre-assignment Details: No participants were excluded
Groups:
- Women With Prolonged Labour: Primi gravidae, single pregnancy, >37 weeks, fetus alive, cephalic presentation.
  Ultrasound examination: Trans-abdominal and trans-perineal 3D ultrasound examination
Period: Overall Study
Arm/Group | Women With Prolonged Labour
Started | 110 (October 2009)
Completed | 110 (August 2010)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Women With Prolonged Labour
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 29 [18 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 0
Region of Enrollment [Number; unit: participants]
  Norway | 110

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Receiver Operating Curve (ROC AUC) Values for Prediction of Vaginal Delivery Using 2D or 3D Ulrasound
Description: Fetal Head descent was first measured as the shortest distance between the outer bony limit of the fetal skull and the Perineum. Fetal head descent was re-assessed by measuring the angle of progression in a mid-sagittal plane. Fetal head-perineum distance was evaluated with using a cut-off of ≤40 mm, while the angle of progression was evaluated using a cut off of ≥ 110 degrees. The ROC curves plotted the percentage sensitivity against the percentage false positive rate for head-perineum distance and angle of progression as measured by ultrasound.
Time Frame: during labor
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Women With Prolonged Labour
Number analyzed (Participants) | 110
percentage probability
  2D fetal head-perineum distance (AUC) | 81 [71 to 91]
  2D angle of progression (AUC) | 76 [66 to 87]
  3D fetal head-perineum distance | 80 [70 to 90]
  3D angle of progression (AUC) | 76 [65 to 86]
Statistical Analysis 1: Comparison: Women With Prolonged Labour; In a previous study we investigated women before induction of labor. Using 40 mm as cut-off level for fetal head - perineum distance, the Cesarean section rate in primiparous women was 7% in the group with a short distance and 27% in the group with a long distance. We assumed similar results, with alpha 0.05, power 0.8 and a ratio of 1 : 1 for the numbers of women with a long and short distance. We would need to include 110 women in the study; Test type: Superiority or Other; p < 0.01, Chi-squared — The reported p-value corresponds with each area under the ROC assessments

2. Secondary Outcome: Percentage of Women With Delivery Within 6 Hours From Defined Prolonged Labor (in Accordance With WHO Recommendations)
Time Frame: 6 hours post determination of prolonged labor
Measure: Number; unit: percentage of participants
Groups:
- Women Delivered Within 6 Hours: Nulliparous women, single pregnancy, > 37 weeks of pregnancy, fetus alive and cephalic presentation.
  Ultrasound examinations: 2D transperineal scan
Arm/Group | Women Delivered Within 6 Hours
Number analyzed (Participants) | 110
percentage of participants
  Fetal head-perineum distance ≤40 mm (n=54) | 74
  Fetal head-perineum distance >40 mm (n=56) | 39
  Angle of progression ≥110 degrees (n=53) | 72
  Angle of progression <110 degrees (n=57) | 44
Statistical Analysis 1: Comparison: Women Delivered Within 6 Hours; Kaplan Meier plots were used to compare time from a defined prolonged labor in the first stage to delivery for 1. women with fetal head-perineum distance ≤40 mm vs. women with distance >40 mm measured with 2D ultrasound. 2. women with angle of progression ≥110 degrees vs. women with angle <110 degrees measured with 2D ultrasound; Test type: Superiority or Other; p < 0.01, Log Rank — the reported p-value corresponds with each log rank comparison

ADVERSE EVENTS:
Time Frame: 1 week
Description: Eventual adverse outcomes were investigated during the postpartum period
Arm/Group | Women With Prolonged Labour
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No